CLINICAL TRIAL: NCT07069283
Title: The Effect of Self-Compassion Practices on Nomophobia Symptoms in Young Adults; A Randomized Controlled Trial
Brief Title: The Effect of Self-Compassion Practices on Nomophobia Symptoms in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Behice Belkıs ÇALIŞKAN, phd, University of Beykent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: E-45778635-050.99-182837
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nomophobia
Keywords: nomophobia symptoms; young adult; self compassion; pain; sleep quality
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal group (Experimental): This group will be given an online self-compassion program for 8 weeks..
  Interventions: Behavioral: Self-Compassion Program
- Control Group (No Intervention): There will be no intervention

INTERVENTIONS:
Behavioral: Self-Compassion Program — Program includes four basic practices: breathing meditation, walking meditation, body scan, and mindful movement. Consciously focusing on what is happening allows people to observe and accept what they are experiencing in their bodies, minds, and the world around them at that moment. Mindfulness practices are an 8-week practice consisting of 2-2.5 hour sessions per week by a trained instructor, mindfulness meditation practices, yoga practices, examining the psychological and physiological aspects of stress, and recently including the concept of self-compassion. In addition, daily practices are given to participants, and a suitable day is determined as a retreat day. The aim is to enable individuals to reveal and experience their thoughts, emotions, and bodily sensations and to increase emotional tolerance by revealing avoidance behaviors. Individuals learn to return to and accept intense bodily sensations and emotional discomfort with mindfulness.
  Arms: Experimantal group

SUMMARY:
The term nomophobia, which can also be defined as a symptom, has emerged with the excessive use of smartphones. Nomophobia is the anxiety and fear that people feel when they are away from their phones for any reason. Nomophobia is defined as the "fear of being deprived of phone or internet access." According to DSM5, "situational phobias are excessive, irrational fears accompanied by anxiety and distress towards a specific object or situation." Considering the anxiety, stress, and worry it creates on individuals, Bragazzi and Del Puente (2014) stated that nomophobia should be added to the DSM-5 due to the dimensions of the anxiety, stress, and worry it creates on individuals and the speed at which it spreads. They explained the symptoms of nomophobia as follows; spending most of the day with a smartphone, constantly checking the battery, in case of being away from the smartphone, thoughts such as the battery or credit running out and not being able to find the phone create anxiety in individuals, staying away from places and spaces where it is not possible to use a smartphone, constantly checking whether notifications or messages have arrived, keeping the smartphone on and nearby even while sleeping, communicating using digital tools because face-to-face conversation creates anxiety, incurring extraordinary expenses for a smartphone or getting into excessive debt.

In addition to making life easier, nomophobia, which occurs with excessive and uncontrolled use of smartphones, can cause some problems. Increasing individuality and the resulting weakening of face-to-face communication bring about addictive applications, depression, headache, visual impairments, sleep problems, musculoskeletal problems, and physiological and psychological problems.

To cope with and manage the symptoms of an addictive condition such as nomophobia, it is envisaged that young adults should be supported with self-compassion practices.

Self-compassion exists from the essence of awareness when we encounter painful and distressing situations. Self-compassion tells individuals to be kind to themselves when they encounter pain and distress. When people encounter an adverse life event, they blame themselves, criticize themselves, react to themselves, and make harmful decisions. A happy and peaceful life emerges thanks to self-compassion, a sense of security, and health. If individuals can accept and tolerate many positive and negative life events and be kind and tolerant towards themselves, they can stop limiting and ignoring their feelings and thoughts. In this way, they can avoid over-identifying by realizing that the experiences experienced are experiences that many people can experience. Individuals with high levels of self-compassion have low levels of depression, anxiety, stress, perfectionism, rumination, and suppressing thoughts. In addition, since they do not judge themselves, their happiness, optimism, enjoyment of life, and motivation are high. In line with this information, self-compassion practices can be supportive during this period when young adults encounter a problem such as nomophobia and have to manage many physiological symptoms. This study aimed to determine the effect of self-compassion practices on nomophobia symptoms in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18-30
* Not having any psychiatric problems

Exclusion Criteria:

* Being under 18 years of age

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-10-28 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Nomophobia Scale | To be filled after the 8-week training program is completed
  File Nomophobia Scale by Yıldırım and Correia (2015) consists of 20 items. The scale is answered from 1 (Strongly Disagree) to 7 (Strongly Agree). The scale is a 7-point Likert type. It consists of 4 sub-dimensions: "Inability to Access Information" (4 items), "Sacrificing Comfort" (5 items), "Inability to Communicate" (6 items) and "Losing Online Connection" (5 items) (Yıldırım and Correia, 2015). Participants are between 20 and 140 on the Nomophobia Scale. It is seen that participants with less than 20 points do not have nomophobia and those with 100-14 points have extreme nomophobia. The original systems of the scale were calculated as .95. The reliability in this study was based on Cronbach's alpha value of .95.

SECONDARY OUTCOMES:
Self-Compassion Scale Short Form (SCF-K) | To be filled after the 8-week training program is completed
  Self-Compassion Scale Short Form (SCF-K); The scale developed by Raes, Pommier, Neff, and Van Gucht (2011) considering it to be more convenient than the long form in terms of time was used. SCF-K, consisting of items taken from the 26-item Self-Compassion Scale, included two items for each subcomponent of self-compassion in order to create this short form, and there are 12 items in total. It is seen that the scale has started to be used in Western literature in recent years, especially due to its ease of use. The Turkish adaptation of the Self-Compassion Scale Short Form was made by Yıldırım and Sarı (2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Beykent ün, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided